CLINICAL TRIAL: NCT01848431
Title: Randomized Study on the Effects of Moderate Anaemia in Free Microvascular Tissue Transfer
Status: Withdrawn | Type: Observational
Why Stopped: staff change and lack of ressources
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: FF-HTC Verson 1-3
Record Dates: First submitted 2013-04-22; First posted 2013-05-07 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2014-12

CONDITIONS: Open Fracture of Foot; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- anaemia group: no blood transfusions will be given until hct falls under 25%
- normal hct group: patients in group 2 will receive transfusions as is currently standard protocol outside the study

SUMMARY:
The evaluation of Perfusion of free flaps in patients with moderate anaemia and possible reduction of the transfusion threshold.

* Trial with surgical intervention

DETAILED DESCRIPTION:
In study group 1 patients will be kept at a hematocrit level below 28% and only receive transfusions if symptomatic or the fall below 25%. Patients in group 2 will receive transfusions to reach a hematocrit always above 30%.

Tissue perfusion in free flaps will be measured with indocyanine green fluorescence angiography, confocal microscopy and oxygen partial pressure measurement probes.

ELIGIBILITY:
Inclusion criteria:

* planned defect reconstruction with free flap and preoperative hematocrit of 28% or below

Exclusion criteria:

* coagulation disorder
* Jehovah's witness
* iodine allergy
* renal or hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for defect reconstruction with free flaps and a preoperative hematocrit of 28 % or below
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Estimated); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of Blood transfusions peri- and postoperative | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, MD, Principal Investigator — University Hospital Zurich, Clinic of Reconstructive Surgery
Locations (1):
- University Hospital Zurich, Center for Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland